CLINICAL TRIAL: NCT03603392
Title: A High-Intensity Exercise Program Stops Weight Regain and Improves Cardiovascular Profile in Post-Bariatric Patients
Brief Title: A High-Intensity Exercise Program in Post-Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Manuel Moya, Principal Investigator, Universidad Miguel Hernandez de Elche
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DPS.MMR.01.15
Record Dates: First submitted 2018-07-04; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Bariatric Surgery and Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: two groups (experimental and control) randomly assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity program (Experimental): Before and after a 5-months of a supervised exercise program were performed in post bariatric patients, body composition, physical fitness and cardiovascular risk factors were measured.
  Interventions: Other: Physical activity program

INTERVENTIONS:
Other: Physical activity program

SUMMARY:
Background: Weight regain is one of the most common problems in bariatric patients. Although exercise contributes to maintaining weight, there are currently few studies performed on this population.

Objective: To know the effects of a high-intensity exercise program applied 3 years after bariatric surgery on body composition and cardiovascular risk factors.

Methods: A 37-month follow-up was performed on 21 patients who underwent bariatric surgery, in which periodic body composition was evaluated. At month 37, participants were divided into an experimental group (EG) and a control group (CG). The EG performed a 5-months of a supervised exercise program. At this point physical fitness, glycemia and cholesterolemia were also evaluated in the EG. Finally, the EG repeated the evaluations 2-months after the end of the program.

DETAILED DESCRIPTION:
A total of 40 patients from the Vinalopó-Salud Hospital of Elche (Spain) who underwent bariatric surgery between 2010-2013, were recruited. Male and female participants were eligible if they complied with the following inclusion criteria: a) absence of cardiovascular disease; b) they had not suffered any type of cancer in the 5-year period before surgery; c) absence of functional limitations that prevented them from performing the exercise program.

Before starting the study, an initial interview was conducted with the patients to verify that they complied with the inclusion criteria. In this interview, all aspects of the program were carefully explained. At the start of the study, all patients who had agreed to participate signed an informed consent. This study was conformed to the Declaration of Helsinki and approved by the Ethics Committees of the University. Two patients declined to participate in the study after the initial interview. Finally, 38 patients started the study and 18 finished it.

One month after surgery, participant's body composition, anthropometric measures and resting blood pressure were assessed. These assessments were performed periodically every six months until month 19 after surgery. At an average of 37.10 ± 4.35 months of follow-up after surgery, they were distributed into two groups, an experimental group (EG; n=10), and a control group (CG; n=8). The EG group performed a monitored exercise program, while only the evaluations were performed in the CG. At this point, measurements of cardiorespiratory fitness and biochemical parameters were added to the previous assessments (anthropometric measures and blood pressure) for the EG. An assessment was performed coinciding with the start of the exercise program (which lasted 20 weeks), and a final assessment was also performed at the end of the program. Finally, the EG was evaluated 2 months after the end of the exercise program.

Body composition, waist and hip circumference, blood pressure and biochemical parameters were evaluated between 8:00 ante meridien (AM) and 9:00 AM. Cardiorespiratory fitness was evaluated between 4:00 post meridien (PM) and 8:00 PM. Measurements were performed in a climatically controlled laboratory, located at 80 m above sea level, in which the relative air humidity was maintained between 45-60% and the temperature between 22-24º.

Body composition, anthropometric measures and cardiovascular risk factors (CVRF) After at least 10 hours of fasting, body composition, biochemical parameters and blood pressure were measured. Alcohol consumption was restricted for at least 8 hours before the test, while PA was forbidden in the 48 hours prior to the test. Participants performed the assessment with an empty bladder. Bioimpedance analysis (Tanita, TBF 300A, Tokyo, Japan) was used to establish body weight and body composition. Body mass index (BMI) was calculated according to the formula: total weight in kilograms divided by squared height in meters (kg·m-2). The International Society for the Advancement of Kinanthropometry (ISAK) protocol was used to assess height and waist and hip circumference. Blood pressure was measured using a digital sphygmomanometer (Microlife WatchBP Home, Heerbrugg, Switzerland), according to established recommendations. Capillary blood samples were taken to analyse blood glucose and Total Cholesterol (TC) using a portable multi-analyser (Accutrend GCT, Roche Diagnostics, Mannheim, Germany).

Cardiorespiratory fitness The peak oxygen uptake (VO2peak) was determined on a cycle ergometer (Technogym Bike Med, Technogym, Gambettola, Italy), using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany) by adapted protocol from Achten. The protocol had two phases: a) a first phase in which the participants performed a 4-minute warm-up at 40 watts (W), followed by increases of 20 W every 3 minutes, maintaining a cadence of 60 rotations per minute (RPM) during the whole phase; and, b) a second phase that started when the respiratory exchange ratio reached 1.0, and which was aimed to determine the VO2peak. This phase consisted of increments of 20 W every minute, maintaining a cadence between 70-80 RPM, until volitional fatigue. The VO2peak was calculated as the average of the highest 30 seconds of VO2. The VO2peak was expressed in absolute values (VO2peak ABS) and normalized to total body weight (VO2peak/BW) and fat-free mass (VO2peak/FFM).

Cardiovascular risk (CVR) The SCORE risk charts of the European Society of Cardiology were used to calculate CVR. The formula to calculate CVR estimates the 10-year coronary risk using TC, systolic blood pressure, gender, age, and smoking status. In addition, CVR was also calculated using waist to hip ratio, and waist to height ratio.

Health-related quality of life The health-related quality of life was measured by the Short Form Health Survey 36 (SF-36), in its version adapted to the Spanish context. This questionnaire measures physical and mental health through 8 scales, the scores of which are transformed to values between 0-100 points, with the highest scores meaning a better function. These 8 scales are grouped into two summary components, the physical summary component, and the mental summary component, which were calculated according to the reference values of the Spanish population, with a mean of 50 and a standard deviation of 10.

The exercise program lasted 20 weeks, which were distributed in five 4-week blocks. The first -block included two weekly sessions, in which the endurance training (ET) and the resistance training (RT) for 5 muscle groups (hamstrings, pectorals, quadriceps, latissimus dorsi, and gastrocnemius) was combined in the same session. In the second block participants trained 3 days a week, in two of them a high-intensity interval training (HIIT) was performed, followed by RT (biceps and triceps were added to the previous 5 major muscle groups trained), while in the third session only the ET was performed. Between the third and fifth block participants trained 4 days a week. In two sessions, a HIIT was performed, followed by RT, focusing on different muscle groups in each session: a) session 1: pectorals, quadriceps, biceps, and hamstrings; b) session 2: dorsal, triceps, gastrocnemius and deltoids. In the other two sessions, ET was performed. In all the blocks, 2 days a week of flexibility training were carried out.

The ET (performed on a cycle-ergometer, elliptical and treadmill) was monitored using a heart rate (HR) monitor (FT40, Polar, Finland). The RT was performed using resistance machines, and training intensity was determined by percentages of 1 maximum repetition which was estimated using the Brzycki formula.

The HIIT consisted of a five-minute warm up, increasing the intensity from 40% of VO2peak to 60% VO2peak. After this, 20 minutes with bouts of 30 seconds at high intensity (60-95% VO2peak) and 30 seconds of active recovery (40% VO2peak), for a total of 10 minutes of training at high intensity were performed. Finally, 3 minutes of cool-down at 40% VO2peak were performed.

ELIGIBILITY:
Inclusion Criteria:

* Absence of cardiovascular disease
* They had not suffered any type of cancer in the 5-year period before surgery
* Absence of functional limitations that prevented them from performing the exercise program

Exclusion Criteria:

-

Ages: 35 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body Composition at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM.
  Body mass index (BMI) was calculated according to the formula: total weight in kilograms divided by squared height in meters (kg·m-2).
  Participants performed the assessment with an empty bladder. Bioimpedance analysis (Tanita, TBF 300A, Tokyo, Japan) was used to establish body weight and body composition.
Change from Baseline waist and hip circumference at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM.
  The ISAK (International Society for the Advancement of Kinanthropometry) protocol was used to assess waist and hip circumference
Change from Baseline Systolic and Diastolic Blood pressure at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM.
  Blood pressure was measured using a digital sphygmomanometer (Microlife WatchBP Home, Heerbrugg, Switzerland), according to established recommendations
Change from Baseline Capillary Blood Samples at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM.. Measurements only performed at the experimental group
  Capillary blood samples were taken to analyse blood glucose and TC using a portable multi-analyser (Accutrend GCT, Roche Diagnostics, Mannheim, Germany)
Change from Baseline Cardiorespiratory Fitness at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM. Measurements only performed at the experimental group
  he peak oxygen uptake (VO2peak) was determined on a cycle ergometer (Technogym Bike Med, Technogym, Gambettola, Italy), using an Oxycon Pro gas analysis system (Jaeger, Friedberg, Germany) by adapted protocol from Achten. The protocol had two phases: a) a first phase in which the participants performed a 4-minute warm-up at 40 watts (W), followed by increases of 20 W every 3 minutes, maintaining a cadence of 60 rotations per minute (RPM) during the whole phase; and, b) a second phase that started when the respiratory exchange ratio reached 1.0, and which was aimed to determine the VO2peak. This phase consisted of increments of 20 W every minute, maintaining a cadence between 70-80 RPM, until volitional fatigue. The VO2peak was calculated as the average of the highest 30 seconds of VO2. The VO2peak was expressed in absolute values (VO2peak ABS) and normalized to total body weight (VO2peak/BW) and fat-free mass (VO2peak/FFM).
Change from Baseline Cardiovascular Risk at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM.
  The SCORE risk charts of the European Society of Cardiology were used to calculate CVR. The formula to calculate CVR estimates the 10-year coronary risk using Total Cholesterol, systolic blood pressure, gender, age, and smoking status. The underlying survival probability, S0, is given by:
  S(age)={S0(age)}exp(w) S(age)={S0(age)}exp(w) S(age+10)={S0(age+10)}exp(w)S(age+10)={S0(age+10)}exp(w) Where w=βchol(cholesterol-6)+βSBP(SBP-120)+βsmoker(current)w=βchol(cholesterol-6)+βSBP(SBP-120)+βsmoker(current)
  For each cause, calculate the 10-year survival probability based on the survival probability for the person's current age and their age in 10 years time:
  S10(age)=S(age+10)/S(age)S10(age)=S(age+10)/S(age) Calculate the 10-year risk for each end-point as Risk10=1-S10(age)Risk10=1-S10(age) The scale range ordered by the 10-year risk of fatal cardiovascular desease are: 15% and over, between 10%-14%, between 5%-9%, Between 3%-4%, 2%, 1%, under 1%.
Change from Baseline Health Status at 5 months | Baseline and 5 months, between 8:00 AM and 9:00 AM. Measurements only performed at the experimental group
  The health-related quality of life was measured by the Short Form Health Survey 36 (SF-36), in its version adapted to the Spanish context. This questionnaire measures physical and mental health through 8 scales, the scores of which are transformed to values between 0-100 points, with the highest scores meaning a better function. These 8 scales are grouped into two summary components, the physical summary component, and the mental summary component, which were calculated according to the reference values of the Spanish population, with a mean of 50 and a standard deviation of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided